CLINICAL TRIAL: NCT06426186
Title: Effect of Right-stellate Ganglion Block in Preventing Postoperative Nausea and Vomiting in Gynecological Laparoscopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PONV-Gynecological surgery
Record Dates: First submitted 2024-04-14; First posted 2024-05-23 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right-stellate ganglion block (Experimental): Right-stellate ganglion block was given 30 minutes before anesthesia induction
  Interventions: Procedure: Right-stellate ganglion block
- Blank control group (No Intervention): No treatment was given 30 minutes before anesthesia induction

INTERVENTIONS:
Procedure: Right-stellate ganglion block — The experimental group was given right stellate ganglion block 30 minutes before anesthesia
  Arms: Right-stellate ganglion block

SUMMARY:
Postoperative nausea and vomiting is one of the common postoperative complications. Studies have reported that without any antiemetic prevention treatment, the overall incidence of PONV in surgical operations is up to 20-30%, and the incidence of PONV in high-risk operations such as gynecological laparoscopy is higher. Postoperative nausea and vomiting can lead to perioperative complications and seriously affect the prognosis of patients. Although various preventive and therapeutic measures have been adopted in clinic, the incidence of perioperative nausea and vomiting is still high. Therefore, it is of great clinical significance to explore more effective and feasible methods to prevent the occurrence of PONV. Stellate ganglion block has been proved to be widely used in clinic and can play a positive role in multiple organs and systems of the whole body. In clinical work, stellate ganglion block is more widely used in the treatment of various pain, autonomic nerve disorders and other diseases. However, there are few clinical studies on whether stellate ganglion block can be used as an effective and feasible means to prevent postoperative nausea and vomiting and the related mechanisms to prevent the possible occurrence of nausea and vomiting. Therefore, this project aims to explore the preventive effect of stellate ganglion block on postoperative nausea and vomiting in gynecological laparoscopic surgery patients, and to explore its possible mechanism.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting is one of the most common postoperative complications second only to postoperative pain. Studies have reported that without any antiemetic prevention treatment, the overall incidence of PONV in surgical operations is up to 20-30%, and the incidence of PONV in high-risk patients such as gynecologic laparoscopy is higher. The pathogenesis of postoperative nausea and vomiting is very complex, including central, peripheral receptors and multiple nerve pathways. When peripheral receptors are stimulated, the signal passes through the afferent nerve to the vomiting center, causing nausea and vomiting. The emetic chemical receptors are rich in many receptors, which can directly feel various toxins, metabolites or drugs in the blood and cerebrospinal fluid, project signals to the nerve center and then spread to the cerebral cortex, causing nausea and vertigo, or transmit signals along the vagus nerve, glossopharyngeal nerve, spinal nerve, etc. to the digestive tract, diaphragm and abdominal wall muscles, resulting in the opening of the sphincter in the upper esophagus and strong contraction of the diaphragm. Abdominal muscles contract, so that the stomach pressure increases, stomach contents through the digestive tract is expelled from the body, vomiting.

There are many factors affecting postoperative nausea and vomiting in gynecological laparoscopic surgery, including patient factors, anesthetic factors and surgical factors. Firstly, gender as an independent risk factor for postoperative nausea and vomiting is widely recognized by researchers, and a large number of studies have confirmed that the incidence of postoperative nausea and vomiting is higher in females, and the possible mechanism is caused by different hormone levels. Secondly, some studies believe that the type of surgery is also a risk factor for postoperative nausea and vomiting, but there is some controversy. In general, laparoscopic surgery patients have a higher incidence of postoperative nausea and vomiting. Finally, the mode of anesthesia and anesthesia-related drugs are also one of the risk factors affecting PONV. Compared with other anesthesia methods, the incidence of PONV was increased under general anesthesia, and the combination of intravenous anesthesia and intraoperative opioid application also increased the incidence of postoperative nausea and vomiting.

Stellate ganglion block has been proved to be widely used in clinic and can play a positive role in multiple organs and systems of the whole body. In clinical work, stellate ganglion block is more widely used in the treatment of various pain, autonomic nerve disorders and other diseases. However, there are few clinical studies on whether stellate ganglion block can be used as an effective and feasible means to prevent postoperative nausea and vomiting and the related mechanisms to prevent the possible occurrence of nausea and vomiting. Therefore, this study will explore the preventive effect of stellate ganglion block on postoperative nausea and vomiting in gynecological laparoscopic patients, and hope to explore its possible mechanism, so as to provide more effective and feasible methods for clinical prevention of postoperative nausea and vomiting and improve patients' medical comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 70 years
2. American Society of Anesthesiologists(ASA) physical status classification I-Ill.
3. Voluntary participation and ability to understand and sign the informed consent form
4. Patients undergoing gynecological laparoscopic surgery elective general anesthesia

Exclusion Criteria:

1. Patients with obesity(BMI>30kg/m2)
2. Contraindicated to stellate ganglion block
3. Patients who cannot cooperate with the study for any reason,or whom the investigator deems unsuitable for inclusion in this trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting | From end of surgery to 24 hours after surgery
  Postoperative nausea and vomiting is evaluated by follow-up

SECONDARY OUTCOMES:
Incidence of nausea and vomiting during preemptive analgesia | From 0-10 minutes after preemptive analgesia
  Postoperative nausea and vomiting is evaluated by investigator's follow-up
Intensity of nausea and vomiting during preemptive analgesia | From 0-10 minutes after preemptive analgesia
  Intensity of nausea and vomiting (the scale is Rhodes index of nausea and vomiting)is evaluated by numerical rating scale (0-10), which higher socre represents more severe the nausea and vomiting
Intensity of nausea and vomiting during hospitalization | From end of surgery to 24 hours after surgery
  Intensity of nausea and vomiting is evaluated by numeric rating scale (0-10), which higher socre represents more uncomfortable
Hemodynamic parameters | When patients enter the operation room (T0),Immediately before intubation（T1，about 30minutes after SGB）,Immediately after intubation（T2，about 35minutes after SGB）， trendelenburg position after completion (T3)，At the end of the operation（T4）
  Mean arterial pressure in mmHg,heart rate in bpm
Postoperative pain intensity | From end of surgery to 24 hours after surgery
  Postoperative pain intensity is assessed by numeric rating scale (0-10), which higher socre represents more uncomfortable
Recovery of gastrointestinal function | From end of surgery to 24 hours after surgery
  Gastrointestinal function is is assessed by the evacuation time
Sleep quality | From end of surgery to 1 day after surgery
  Sleep quality is is assessed by numeric rating scale (0-10), which higher socre represents better sleep quality
Satisfaction score and postoperative analgesia satisfaction score | From end of surgery to hospital discharge with about 5 days
  Satisfaction score and postoperative analgesia satisfaction score is assessed by numeric rating scale (0-10), which higher socre represents more comfortable

CONTACTS AND LOCATIONS:
Overall Officials: ling Dan, BD, Principal Investigator — The Second Affilated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication

REFERENCES:
- [Derived] Liu Y, Piao G, Chen J, Duan G, Dan L, Chen G, Zhang Y. Effect of Right Stellate Ganglion Block on Preventing Postoperative Nausea and Vomiting in Gynecological Laparoscopic Patients: A Randomized Controlled Trial. Adv Ther. 2025 Mar;42(3):1537-1549. doi: 10.1007/s12325-025-03109-7. Epub 2025 Feb 10. PMID 39928244